CLINICAL TRIAL: NCT03125070
Title: INSPIRE: A Multicenter Randomized Controlled Trial Integrating Health Informatics in a Scalable Stepped Care Self-Management Program for Survivors After Hematopoietic Cell Transplantation
Brief Title: Self-Management Program and Survivorship Care Plan in Improving the Health of Cancer Survivors After Stem Cell Transplant
Acronym: INSPIRE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, K. Scott Baker, Professor, Fred Hutchinson Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 9819; NCI-2017-00583 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9819 (Other: Fred Hutch/University of Washington Cancer Consortium); R01CA215134 (NIH); RG1001537 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2017-04-19; First posted 2017-04-24 (Actual); Results first posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (INSPIRE, survivorship care plan) (Experimental): Patients receive immediate access to the INSPIRE online program and personalized survivorship care plan.
  Interventions: Other: Internet, Mobile app and Telehealth Intervention; Other: Survey Administration
- Group II (usual care) (Active Comparator): Patients receive an online program linking to existing online survivor resources and a personalized survivorship care plan. Patients may receive access to the INSPIRE online program after 12 months.
  Interventions: Other: Best Practice and Internet site with links to existing resources; Other: Survey Administration

INTERVENTIONS:
Other: Best Practice and Internet site with links to existing resources — Receive usual care
  Other Names: best practice; standard of care; standard therapy
  Arms: Group II (usual care)
Other: Internet, Mobile app and Telehealth Intervention — Receive INSPIRE and survivorship care plan
  Other Names: Digital Intervention
  Arms: Group I (INSPIRE, survivorship care plan)
Other: Survey Administration — Ancillary studies

SUMMARY:
This phase III trial investigates health informatics and a self-management program for improving the health of cancer survivors after stem cell transplant. After transplant many survivors may feel stressed or may be unsure of what health care they need. A self-management program called "INSPIRE," along with a personalized survivorship care plan may improve stress and health care for transplant survivors.

DETAILED DESCRIPTION:
OUTLINE:

Patients are randomized to 1 of 2 groups.

GROUP I: Patients receive immediate access to the INSPIRE online program and personalized survivorship care plan.

GROUP II: Patients receive an online program linking to existing online survivor resources and a personalized survivorship care plan. Patients receive access to the INSPIRE online program after 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Received >= 1 autologous or allogeneic (related or unrelated) HCT with curative intent at a participating transplant center for a hematologic malignancy
* Age 18 years of age or older at last transplant
* Survival 2-5 years after last HCT when first approached for enrollment
* In remission at time of study entry, may be receiving chemoprevention
* Internet and email access
* American and Canadian citizens, and/or those with mailing addresses in the United States (US)/Canada and/or temporarily residing anywhere outside the country (IE - military).

Exclusion Criteria:

* Development of invasive subsequent malignancy after HCT other than non-melanoma skin cancer, in the past two years
* Medical or other issue prohibiting computer use, reading or ability to comply with all study procedures or unable to communicate via phone (e.g., significant vision, hearing or cognitive impairment, major illness, hospitalization)
* Residing in an institution or other living situation where health care decisions are not made by the participant (e.g., hospitalized, prisoners, living in a rehabilitation facility)
* Does not complete baseline patient-reported outcome (PRO) assessment items required to determine stratification or whether the survivor meets inclusion and exclusion criteria
* Non-proficient in English (written and spoken)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 546 (Actual)
Dates: Start 2020-10-29 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: K. Scott Baker, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (15):
- United States (15):
  - Moffitt Cancer Center, Tampa, Florida
  - Loyola University Medical Center, Maywood, Illinois
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - National Marrow Donor Program, Minneapolis, Minnesota
  - Center for International Blood and Marrow Transplant Research, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Roswell Park Cancer Institute, Buffalo, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Texas Oncology at Baylor Charles A Sammons Cancer Center, Dallas, Texas
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Number analyzed excludes 34 participants determined to be ineligible after consent and 137 participants identified as not requiring the intervention due to lack of distress and adherence to healthcare screening reccomendations.
  This leaves 375 participants included in the final analyses.
Period: Overall Study
Arm/Group | Group I (INSPIRE, Survivorship Care Plan) | Group II (Usual Care)
Started | 184 | 191
Completed | 129 | 159
Not Completed | 55 | 32

BASELINE CHARACTERISTICS:
Population: Number analyzed excludes 34 participants determined to be ineligible after consent and 137 participants identified as not requiring the intervention due to lack of distress and adherence to healthcare screening reccomendations.
  This leaves 375 participants included in the final analyses.
Groups:
- Group I (INSPIRE, Survivorship Care Plan): Participants receive immediate access to the INSPIRE online program and personalized survivorship care plan.
  Internet, Mobile app and Telehealth Intervention: Receive INSPIRE and survivorship care plan
  Survey Administration: Ancillary studies
- Group II (Usual Care): Participants receive an online program linking to existing online survivor resources and a personalized survivorship care plan. Participants may receive access to the INSPIRE online program after 12 months.
  Best Practice and Internet site with links to existing resources: Receive usual care
  Survey Administration: Ancillary studies
- Total: Total of all reporting groups
Arm/Group | Group I (INSPIRE, Survivorship Care Plan) | Group II (Usual Care) | Total
Number analyzed (Participants) | 184 | 191 | 375
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 117 | 132 | 249
  >=65 years | 67 | 59 | 126
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.11 (12.8) | 57.3 (12.5) | 58.2 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 99 | 184
  Male | 99 | 92 | 191
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 8
  Not Hispanic or Latino | 177 | 186 | 363
  Unknown or Not Reported | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 4 | 4 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 5 | 11 | 16
  White | 167 | 163 | 330
  More than one race | 2 | 6 | 8
  Unknown or Not Reported | 5 | 4 | 9
Region of Enrollment [Number; unit: participants]
  United States | 181 | 190 | 371
  Canada | 3 | 1 | 4
Cancer and Treatment Distress [Count of Participants; unit: Participants] — The CTXD is a 22-item inventory of distress or worry related to stressful events for cancer survivors.The count of participants reported is the number of participants who reported distress or worry at baseline.
  Participants | 77 | 93 | 170
Healthcare Adherence (HCA) [Count of Participants; unit: Participants] — The HCA is derived from the Cornell Service Index. Scores are transformed to proportion of HCA recommendations met. For primary outcomes, we use HCA items reflecting adherence to cardiometabolic surveillance (HCA-CM; 5 items). The count of participants reported is the number of participants that did not meet cardiovascular surveillance reccomendations at baseline.
  Participants | 95 | 114 | 209

OUTCOME MEASURES:

1. Primary Outcome: Cancer and Treatment Distress (CTXD)
Description: Among those impaired at baseline, percent who are no longer impaired at 12 months (among those not missing either). Scores range from 0-3 and higher scores indicate higher distress. A cutoff of >=.90 was used to categorize participants as high in distress. Participants with scores <.90 were categorized as not distressed.
Time Frame: Up to 12 months
Population: Group that met criterion for highly distressed
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group I (INSPIRE, Survivorship Care Plan) | Group II (Usual Care)
Number analyzed (Participants) | 77 | 93
percentage of participants | 23.4 [14.5 to 34.4] | 22.6 [14.6 to 32.4]
Statistical Analysis 1: Comparison: Group I (INSPIRE, Survivorship Care Plan) vs Group II (Usual Care); Test type: Superiority; p = 0.90, Chi-squared — The threshold for statistical significance was p=0.05

2. Primary Outcome: Health Care Adherence (HCA)-Cardiometabolic
Description: Assesses adherence to cardiometabolic surveillance in intervention participants vs. controls. Among those impaired at baseline, percent no longer impaired at 12 months. Scores range from 0-1. Higher scores indicate high adherence. A cutoff of <.80 was used to categorize participants as low in adherence. Scores higher than .80 were classified as being adherent to cardiometabolic surveillance.
Time Frame: Up to 12 months
Population: Those impaired at baseline
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group I (INSPIRE, Survivorship Care Plan) | Group II (Usual Care)
Number analyzed (Participants) | 95 | 114
percentage of participants | 30.5 [21.5 to 40.8] | 27.2 [19.3 to 36.3]
Statistical Analysis 1: Comparison: Group I (INSPIRE, Survivorship Care Plan) vs Group II (Usual Care); Test type: Superiority; p = 0.60, Chi-squared — The threshold for statistical significance was p=0.05

3. Primary Outcome: Characteristics of Intervention Participants Who Require Telehealth Stepped Care at 6-weeks
Description: Determine characteristics of participants who 1) do not meet criteria for adequate knowledge of cardiometabolic risks, or 2) do not report improved distress, or 3) have not logged in to the online program.
Time Frame: 6-weeks after enrollment.
Population: Intervention participants who require telehealth stepped care at 6-weeks
Measure: Count of Participants; unit: Participants
Groups:
- Telehealth-Yes: Intervention participants who required telehealth stepped care
- Telehealth-No: Intervention participants who did not require telehealth stepped care
Arm/Group | Telehealth-Yes | Telehealth-No
Number analyzed (Participants) | 68 | 116
Participants
  Sex-Female | 35 | 50
  Sex-Male | 33 | 66
  Age at baseline <70 | 54 | 91
  Age at baseline >=70 | 14 | 25
  White/non-Hispanic | 61 | 103
  BIPOC | 6 | 10
  Race/ethnicity unknown | 1 | 3
  Education: High school diploma or less | 6 | 18
  Education: At least some college or vocational/technical program | 62 | 97
  Education level unknown | 0 | 1
  Income: <$100,000 | 39 | 75
  Income: >=$100,000 | 26 | 34
  Income unknown | 3 | 7
  PHQ score <10 (no depression) | 56 | 98
  PHQ 10-14 (mild depression) | 6 | 13
  PHQ 15-19 (moderate depression) | 5 | 2
  PHQ >=20 (severe depression) | 1 | 2
  PHQ score unknown | 0 | 1
  CTXD <0.9 (not distressed) | 26 | 52
  CTXD >=0.9 (distressed) | 42 | 62
  CTXD score unknown | 0 | 2
  HCU-C >.80 (normal adherence) | 13 | 35
  HCU-C <.80 (low adherence) | 53 | 78
  HCU-C unknown | 2 | 3
  HCU-SM >=.80 (normal adherence) | 45 | 85
  HCU-SM <.80 (low adherence) | 23 | 31
Statistical Analysis 1: Comparison: Telehealth-Yes vs Telehealth-No; Sex: Female vs. Male; Test type: Other; p = 0.27, Chi-squared — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Telehealth-Yes vs Telehealth-No; Age <70 vs. >=70; Test type: Other; p = 0.88, Chi-squared — The threshold for statistical significance was p=0.05
Statistical Analysis 3: Comparison: Telehealth-Yes vs Telehealth-No; Race and ethnicity: white AND non-Hispanic versus any other combination of race and ethnicity (BIPOC); Test type: Other; p = 0.98, Chi-squared — The threshold for statistical significance was p=0.05; Participants that did not answer this survey item are shown as unknwon in the table and are excluded from the statistical test
Statistical Analysis 4: Comparison: Telehealth-Yes vs Telehealth-No; Education: High school or less versus at least some college or vocational/technical program; Test type: Other; p = 0.19, Chi-squared — The threshold for statistical significance was p=0.05; [statistical method as in outcome 3, analysis 3]
Statistical Analysis 5: Comparison: Telehealth-Yes vs Telehealth-No; Income: <$100,000 annual versus >=$100,000 annual; Test type: Other; p = 0.24, Chi-squared — The threshold for statistical significance was p=0.05; [statistical method as in outcome 3, analysis 3]
Statistical Analysis 6: Comparison: Telehealth-Yes vs Telehealth-No; PHQ score at baseline: no depression (<10), mild depression (10-14), moderate depression (15-19), severe depression (>=20); Test type: Other; p = 0.28, Chi-squared — The threshold for statistical significance was p=0.05; Participants that did not answer the survey items for this measure are shown as unknwon in the table and are excluded from the statistical test
Statistical Analysis 7: Comparison: Telehealth-Yes vs Telehealth-No; CTXD score at baseline <0.9 (not distressed) or >=0.9 (distressed); Test type: Other; p = 0.33, Chi-squared — The threshold for statistical significance was p=0.05; [statistical method as in outcome 3, analysis 6]
Statistical Analysis 8: Comparison: Telehealth-Yes vs Telehealth-No; Cardiometabolic Healthcare Utilization (HCU-C) score at baseline: >.80 versus <.80; Test type: Other; p = 0.10, Chi-squared — The threshold for statistical significance was p=0.05; [statistical method as in outcome 3, analysis 3]
Statistical Analysis 9: Comparison: Telehealth-Yes vs Telehealth-No; Secondary cancer screening healthcare utilization (HCU-SM) at baseline: >=.80 versus <.80; Test type: Other; p = 0.31, Chi-squared — The threshold for statistical significance was p=0.05

4. Secondary Outcome: Health Care Adherence (HCA)-Subsequent Malignancy Screening
Description: Assesses adherence to subsequent malignancy surveillance in intervention participants vs. controls. Among those impaired at baseline, percent no longer impaired at 12 months.
Time Frame: Up to 12 months
Population: Participants impaired at baseline
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group I (INSPIRE, Survivorship Care Plan) | Group II (Usual Care)
Number analyzed (Participants) | 42 | 48
percentage of participants | 4.8 [0.6 to 16.2] | 4.2 [0.5 to 14.3]
Statistical Analysis 1: Comparison: Group I (INSPIRE, Survivorship Care Plan) vs Group II (Usual Care); Test type: Superiority; p = 0.89, Chi-squared

5. Secondary Outcome: PHQ-8 Depression
Description: Assessed by participant questionnaire.Among those impaired (PHQ≥10) at baseline, percent no longer impaired at 12 months
Time Frame: Up to 12 months
Population: Participants impaired at baseline
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group I (INSPIRE, Survivorship Care Plan) | Group II (Usual Care)
Number analyzed (Participants) | 21 | 38
percentage of participants | 28.6 [11.3 to 52.2] | 39.5 [24.0 to 56.5]
Statistical Analysis 1: Comparison: Group I (INSPIRE, Survivorship Care Plan) vs Group II (Usual Care); Test type: Superiority; p = 0.40, Chi-squared

6. Other Pre Specified Outcome: Knowledge of Survivorship Needs and Health Related Self-efficacy
Description: Mediators of primary outcomes: assessed by patient questionnaires.
Time Frame: Up to 12 months
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Reach, Engagement and Fidelity of Web-based Intervention
Description: Process Measures: Rates of participants approached versus registering, rates of visits to the web site, pages viewed, types of modalities used, attrition rates and support requests.
Time Frame: Up to 12 months
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Cost and Resources to Maintain Program
Description: Determine resources that would be needed to sustain the intervention as a national HCT survivorship program if implemented through the CIBMTR/NMDP.
Time Frame: 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year
Description: This clinical trial is a behavioral intervention.
Arm/Group | Group I (INSPIRE, Survivorship Care Plan) | Group II (Usual Care)
All-Cause Mortality (participants affected / at risk) | 3/184 | 1/191
Serious Adverse Events (participants affected / at risk) | 0/184 | 0/191
Other Adverse Events (participants affected / at risk) | 0/184 | 0/191

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-28): https://cdn.clinicaltrials.gov/large-docs/70/NCT03125070/Prot_SAP_000.pdf